CLINICAL TRIAL: NCT00363285
Title: Intermittent Hormone Therapy for Newly Diagnosed Metastatic Prostate Cancer
Brief Title: Cyproterone Acetate in Treating Patients With Newly Diagnosed Stage III or Stage IV Prostate Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Bartholomew's Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000495321; SEUG-9901; BARTS-SEUK-9901; MREC-04/5/006; BARTS-P/02/203; EU-20630
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2006-10

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gonadotropin-Releasing Hormone; Cyproterone Acetate

INTERVENTIONS:
Biological: gonadotrophin releasing hormone
Drug: cyproterone acetate
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Hormone therapy, such as cyproterone acetate may stop the adrenal glands from making androgens. Sometimes the tumor may not need treatment until it progresses. In this case, observation may be sufficient. It is not yet known whether giving cyproterone acetate continuously is more effective than giving cyproterone acetate after tumor progression in treating prostate cancer.

PURPOSE: This randomized phase III trial is studying cyproterone acetate to compare how well it works when given continuously or after tumor progression in treating patients with newly diagnosed stage III or stage IV prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare time to loss of androgen dependence, based on serum prostate-specific antigen failure, in patients with newly diagnosed stage III or IV prostate cancer treated with intermittent vs continuous androgen suppression comprising cyproterone acetate.
* Compare time to treatment failure (subjective or objective progression) in patients treated with these regimens.
* Compare quality of life of patients treated with these regimens.
* Compare survival of patients treated with these regimens.

Secondary

* Compare the side effects in patients treated with these regimens.
* Determine the first and total therapy-free intervals in patients treated with intermittent cyproterone acetate.

OUTLINE: This is a randomized, multicenter study.

All patients receive cyproterone acetate daily for 16 weeks. Patients also receive monthly injections of luteinizing hormone-releasing hormone (LHRH) agonist beginning in week 2 and continuing for 14 weeks. Patients with a prostate-specific antigen (PSA) level of ≤ 4 ng/mL and who are asymptomatic at 14 weeks are randomized to 1 of 2 treatment arms.

* Arm I (continuous maximum-androgen blockade): Patients receive cyproterone acetate daily and monthly LHRH agonist depot injections in the absence of disease progression or unacceptable toxicity. Patients may also undergo orchidectomy.

Quality of life is assessed every 6 months for 2 years and then annually thereafter.

* Arm II (intermittent treatment): Patients are observed after randomization. Treatment with daily cyproterone acetate resumes if symptoms demand hormone treatment and patient has any PSA level OR if patient is asymptomatic and has a PSA level ≥ 20 ng/mL. Treatment continues in the absence of disease progression or unacceptable toxicity. If after 9 months of treatment, a PSA level of ≤ 4 ng/mL is not achieved or the patient remains symptomatic, treatment is discontinued.

Quality of life is assessed every 6 months and when therapy is restarted.

Pain and performance status are assessed at each visit in both treatment arms.

After completion of study therapy, patients are followed periodically.

PROJECTED ACCRUAL: A total of 900 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * T3 -T4, M0-M1 (stage III or IV disease)
* Prostate-specific antigen level ≥ 4 ng/mL and ≤ 100 ng/mL

PATIENT CHARACTERISTICS:

* Performance status 0-2
* Normal liver function
* No other neoplasia (except skin, excluding melanoma)
* No expected difficulties of follow-up related to psychiatric disorders, marked senility, or too large a distance between patient's home and investigator's center
* No severe chronic disease

PRIOR CONCURRENT THERAPY:

* No prior hormonal therapy or chemotherapy
* No prior surgery (radical prostatectomy), except transurethral resection, for M0 patients
* No prior radiotherapy to the primary tumor for M0 patients

Max Age: 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2003-01

PRIMARY OUTCOMES:
Time to loss of androgen-dependence, based on serum prostate-specific antigen (PSA) failure according to protocol definition
Time to treatment failure (subjective or objective progression)
Quality of life
Survival

SECONDARY OUTCOMES:
Side effects
First and total therapy-free intervals in patients treated with intermittent cyproterone acetate

CONTACTS AND LOCATIONS:
Overall Officials: R. T. Oliver, MD, Study Chair — St. Bartholomew's Hospital
Locations (2):
- United Kingdom (2):
  - Saint Bartholomew's Hospital, London, England
  - Scarborough General Hospital, Scarborough, England